CLINICAL TRIAL: NCT01002937
Title: Novel Prognostic Markers in Renal Cancer: a Protocol for the Analysis of Paraffin Embedded Tumour Samples
Brief Title: Novel Prognostic Markers in Renal Cancer
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, RMH R&D, Professor Martin Gore, Royal Marsden NHS Foundation Trust
Other Study IDs: CCR3076
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Renal Cell Carcinoma
Keywords: Biomarkers; Prognosis response to treatment; Renal cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tumour tissue, renal cell carcinoma: > 2mm x 2mm of tumour tissue obtained from paraffin blocks taken from biopsies or nephrectomy specimens.

SUMMARY:
The purpose of this project is to analyze tumour tissue from a group of subjects with renal cell carcinoma, who have been treated at the Royal Marsden Hospital.

DETAILED DESCRIPTION:
Renal cancers have different clinical outcomes. The principal research objective is to study tumour tissue from renal cancer patients and try and understand why some cancers progress more rapidly than others. Further, another key aim of this study is to try and understand why some patients respond to treatment and others do not.

ELIGIBILITY:
Inclusion Criteria:

* The presence of histologically proven renal cell cancer
* The availability of paraffin embedded tissue
* Informed consent needed for tissue taken after January 2006 (date of enforcement of human tissue act)

Exclusion Criteria:

* Absence of histological tissue
* Absence of consent to study tissue after January 2006

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Tumour tissue from subjects with renal cell carcinoma, who have been treated at the Royal Marsden Hospital
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2008-12-01 (Actual); Primary Completion 2014-12-17 (Actual); Study Completion 2014-12-17 (Actual)

PRIMARY OUTCOMES:
The profiling of the expression of signal transduction biomarkers, gene expression, gene copy numbers and effect of mutations of the VHL gene in renal cancer and their relationship to clinical outcomes. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Professor Martin Gore, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom